CLINICAL TRIAL: NCT04744558
Title: Effects of Calorie Restricted Low Carbohydrate High Fat Ketogenic vs. Non-ketogenic Diet on Strength, Body Composition, Hormonal and Lipid Profile in Trained Middle-aged Men
Brief Title: Low Carbohydrate High Fat Ketogenic vs. Non-ketogenic Diet
Acronym: LCHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Vladimir Vidic, MSc, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 484-2
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Ketogenic Dieting
Keywords: Ketogenic diet; Testosterone; Insulin; Body-composition; Resistance-training; Middle-aged men
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic (Experimental): Low carb high fat ketogenic diet
  Interventions: Other: Low carb high fat ketogenic dieting
- Non-ketogenic (Active Comparator): Low carb high fat non-ketogenic diet
  Interventions: Other: Low carb high fat non-ketogenic dieting

INTERVENTIONS:
Other: Low carb high fat ketogenic dieting — Macronutrient ratios for low carb high fat ketogenic diet were 20 %, 5 %, 75 % of protein, carbohydrates and fat, respectively. Caloric intake for experimental phase was set to cover basal metabolism and sedentary activities (BMR times 1.2) for every participant using the Mifflin St Jeor equation.
  Arms: Ketogenic
Other: Low carb high fat non-ketogenic dieting — Macronutrient ratios for low carb high fat non-ketogenic diet were 20 %, 15 %, 65 % of protein, carbohydrates and fat, respectively. Caloric intake for experimental phase was set to cover basal metabolism and sedentary activities (BMR times 1.2) for every participant using the Mifflin St Jeor equation.
  Arms: Non-ketogenic

SUMMARY:
The aim of this paper was to investigate and compare the effects of two iso-energetic hypo-caloric ketogenic hyper-ketonemic and non-ketogenic low carbohydrate high fat high cholesterol diets on body-composition, muscle strength and hormonal profile in experienced resistance-trained middle-aged men. Twenty non-competitive experienced resistance-trained middle-aged men were on the supervised calorie maintenance western diet and resistance-training regimen for 4 weeks and then divided into ketogenic and non-ketogenic groups for 8 weeks period. Keto bodies (β-hydroxybutyrate) levels were measured weekly, testosterone and insulin biweekly, strength and body-composition monthly, lipid profile and blood sugar level at the beginning and at the end of the study.

DETAILED DESCRIPTION:
The primary goal of this research was to investigate and compare the effects of two forms of hypo-caloric LCHF high cholesterol ketogenic hyper-ketonemic and non-ketogenic diets on muscle strength and body-composition in the experienced resistance-trained middle-aged healthy male population, and explore possible advantage of ketogenic state. The secondary goal was to examine the rate and magnitude of hormonal changes during the 8 weeks dietary phase and their possible impact on the muscle strength and body-composition. It is hypothesized that calorie intake is the main variable that influences body-compositional changes regardless of the ketogenic state in similar LCHF dieting conditions.

Four weeks before the experimental procedure participants undertook a detailed medical examination and subsequently were familiarized with all testing schedules and new training facilities in which they continued supervised training sessions, with equalized exercise selection and order for every muscle group as well as for volume and intensity. Participants were instructed not to change any of their current eating habits supervised for the total energy intake set at the calorie maintenance requirement, until the beginning of the LCHF dietary phase of the experiment. After completing 4 weeks of the familiarization phase, the subjects were randomized into ketogenic (KG) and non-ketogenic group (NKG). The first group received LCHF high-cholesterol ketogenic dietary treatment, and the second group received LCHF high-cholesterol non-ketogenic dietary treatment, with the equally reduced calorie intake. The experimental dietary phase lasted for 8 weeks without any change in resistance training.

Blood ketones were monitored weekly, hormonal values every 2 weeks, muscle strength and body-composition every 4 weeks, and basic blood analysis with lipid profile and blood sugar level at the beginning and at the end of the dietary phase of the study Twenty healthy non-competitive experienced resistance-trained middle-aged men (Age = 42.7±1.5 years, Body height = 181.7±4.6 cm, Body mass (BM) = 88.3±5.8 kg), without any recent medical condition, were selected for this research. Inclusion criteria were more than 5 years of experience with resistance-training, and a minimum of 2 years of training continuity prior to the study, with one repetition maximum (1RM) lower limit for bench press at 100% body weight and for squat at 130% bodyweight. In addition, including criteria pertaining to dietary habits, was that no major change in nutrition regime (prolonged increase or decrease in calories or a macronutrient percentage change) was taken in the last 6 months prior to the study. No recent injuries and no medical treatment were mandatory conditions for participation in the study. After initial consultations, participants were asked to avoid alcohol and training stimulants. All participants gave written informed consent for study protocol, approved by the Ethical committee of the Faculty of Sport and Physical Education (IRB: 484-2).

The training was conducted in the same sports facility, supervised by qualified certified professionals at the same time of the day, with the beginning between 18 h and 19 h, four times per week on working days. After initial strength testing 4 weeks prior to the dietary change, subjects training was equalized by the exercise selection, training volume, and intensity based on their individual 1RM. Every major muscle group was trained twice per week with free weights and auxiliary cable exercises in the 6 - 12 repetitions range and 60 - 90 seconds between sets and 2 - 3 minutes between exercises. If any of the subjects missed the training session it was allowed to complete it on another day of the week. Missing training completely meant disqualification from the study. All participants were instructed not to perform any additional physical exercise of any type during the study.

At the beginning of the experimental phase, which followed supervised lead-in calorie maintenance habitual diet phase, weekly LCHF ketogenic and non-ketogenic meal plans were given to the participants with the additional individual verbal instructions. All supervision and guidance were carried through on a weekly base by registered dietitian. Collective supervised attainment of the food supply for every next week was conducted from the same supermarket brand in 2 locations. Additional individual consultations, if needed, were provided for all participants at any time point throughout the study, ensuring compliance to the diet. Every participant was provided with the calibrated kitchen scale (Profi Cook PC-KW 1061) for the duration of the experiment. LCHF diet consisted mainly of meat (beef and veal, poultry), fish (salmon, sardines, tuna), butter and coconut oil for cooking, fat cheese, flaxseed and olive oil for salad dressing and green vegetables. Whole eggs were mandatory on the daily basis insuring intended adequate cholesterol intake. The NKG group obtained their additional small amount of carbohydrate intake from brown rice. Protein intake was set to be equal for both experimental groups with differences in CHO and fat content. Macronutrient ratios for KG and NKG groups were set to 20 %, 5 %, 75 % vs. 20 %, 15 %, 65 % of protein, carbohydrates and fat, respectively. Caloric intake for experimental phase was set to cover basal metabolism and sedentary activities (BMR times 1.2) for every participant using the Mifflin St Jeor equation providing that energy deficit comes primarily from training activities. Dietary intake was calculated using the Diet Master Pro 14.4 software.

All participants were monitored weekly to achieve and sustain blood β-hydroxybutyrate (BHB) level of 1 mmol and above in KG and limit it to 0.1 - 0.2 mmol levels in NKG, throughout the whole duration of the study. If any of the participants were to cross the marked values of the BHB levels in either direction, evaluation and correction of CHO intake would have been immediately carried through, and remeasuring was scheduled before the next training session.

All the biochemical testing, except blood ketone values (BHB), were done on Sunday mornings after a complete day of rest from the last training session on Friday's. Blood samples were obtained via venipuncture by trained phlebotomists in the morning at 08 h after 12 hours fast to avoid diurnal variations. Whole blood was collected, transferred into appropriate tubes for obtaining serum and plasma, and subsequently centrifuged at 1,500 g for 15 min at 4°C. Resulting serum and plasma were stored at -80°C until analysis which was done on the Roche Hitachi Cobas c 311 and c 411 (Roche Diagnostics, Hitachi, Tokyo, Japan) using ECLIA and Spectrophotometry methods for testing testosterone, insulin, blood lipid levels (Total cholesterol, High density lipoprotein, Low density lipoprotein, Triglycerides) and blood glucose levels, while ELISA reader RAYTO RT-2100C (Pioway Medical Lab Equipment, Nanjing, China) was used for determining free testosterone levels. All hormones were measured in the same assay in duplicate measurements on the same day to avoid compounded inter-assay variance. The norm for validity of the measurements was intra-assay variance set to less than 5% for all analyses.

The BHB samples were taken from the finger blood sample, using a Precision Xtra™ meter (Abbott Diabetes Care, Alameda, CA) and were measured in the late afternoon between 17 h and 18 h, before collective training. This timing was chosen as optimal to avoid possible misreading due to the morning cortisol and training influence.

Maximal strength was determined via 1RM bench press (BP) and squat (SQ) measurements in accordance with International Powerlifting Federation rules. After performing general (stationary bicycle) and specific (sets with 50% and 75% of predicted 1RM) warm up, subjects had up to 5 attempts to achieve 1RM. Every attempt was accompanied by strong verbal encouragement. All testing was done at the same time of day in which subjects had their training sessions after two days of rest from the last training.

Body-composition parameters, lean body mass (LBM) and fat mass (FM) were obtained in the morning after an overnight fast on empty stomach using an electric scale, bio-impedance device (In Body 720; Biospace Co., Soul, Korea) using the standardized procedure recommended by the manufacturer and previous studies. In brief, participants were in a standing position with hands and feet placed on the electrodes. Testing was done and monitored by qualified laboratory personnel. Participants were instructed to come without any physical effort prior to the testing.

All measurements and testing were done in accordance with Helsinki declaration and rules of the Ethic Committee of the Faculty of Sport and Physical Education.

Basic descriptive statistic (Mean, SD) was performed, following a visual inspection of boxplots for identifying outliers. Normality test was performed for confirmation of the normality of the data. T test was used to identify differences between lead in and experimental diets. Mixed (split plot) ANOVA was used to determine the time, group, and treatment x time interactions. When a significant F-value was found, post-hoc with Bonferroni adjustment was used for multiple comparisons. Data were reported as mean ± standard deviation. The level of significance was set at p < 0.05. The program used for statistical analysis was SPSS 19 (IBM).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were more than 5 years of experience with resistance-training, and a minimum of 2 years of training continuity prior to the study, with one repetition maximum (1RM) lower limit for bench press at 100% body weight and for squat at 130% bodyweight. In addition, including criteria pertaining to dietary habits, was that no major change in nutrition regime (prolonged increase or decrease in calories or a macronutrient percentage change) was taken in the last 6 months prior to the study. No recent injuries and no medical treatment were mandatory conditions for participation in the study.

Exclusion Criteria:

* Noncompliance to the diet, and the missing training schedule.

Ages: 40 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study focused on strength-trained middle-aged men
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Hormonal changes | 8 weeks
  Testosterone, free testosterone and insulin assessment

SECONDARY OUTCOMES:
Body composition changes | 8 weeks
  Lean body mass and fat free mass assessment
Muscle strength changes | 8 weeks
  Muscle strength assessment

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir M Vidić, MSc, Principal Investigator — Faculty of Sport and Physical Education, University of Belgrade
Locations (1):
- Faculty of Sport and Physical Education, Belgrade, Serbia